CLINICAL TRIAL: NCT02719808
Title: A Cohort Study of Tenofovir on Blocking HBV Intrauterine Infection
Brief Title: Study of Antiretroviral Therapy to Prevent HBV Intrauterine Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AHCR2014-018
Record Dates: First submitted 2016-03-06; First posted 2016-03-25 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Hepatitis B, Chronic
Keywords: Vertical infection transmission; Tenofovir
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, placenta tissue of HBeAg-positive pregnant women
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Tenofovir1: 100 patients receive tenofovir （300mg/d）from (28±2） weeks of pregnancy to one week after delivery.
  Interventions: Drug: Tenofovir1
- Tenofovir2: 100 patients receive tenofovir （300mg/d）from (28±2） weeks of pregnancy to one month after delivery.
  Interventions: Drug: Tenofovir2
- Tenofovir3: 100 patients receive tenofovir （300mg/d）from （24±2）weeks of pregnancy to one week after delivery.
  Interventions: Drug: Tenofovir3
- Tenofovir4: 100 patients receive tenofovir （300mg/d）from （24±2）weeks of pregnancy to one month after delivery.
  Interventions: Drug: Tenofovir4
- Group without any treatment: 100 patients don't receive any blockade therapies

INTERVENTIONS:
Drug: Tenofovir1 — receive tenofovir （300mg/d）from （28±2）weeks of pregnancy to one month after delivery, it is the observational exposure.
  Groups: Tenofovir1
Drug: Tenofovir2 — receive tenofovir （300mg/d）from（28±2）weeks of pregnancy to one month after delivery, it is the observational exposure.
  Groups: Tenofovir2
Drug: Tenofovir3 — receive tenofovir （300mg/d）from （20±2）weeks of pregnancy to one month after delivery, it is the observational exposure.
  Groups: Tenofovir3
Drug: Tenofovir4 — receive tenofovir （300mg/d）from （20±2）weeks of pregnancy to one week after delivery, it is the observational exposure.
  Groups: Tenofovir4

SUMMARY:
500 pregnant patients with HBeAg-positive and HBV-DNA≥ 106copies /ml who will do their pregnant check in the First Affiliated Hospital of Xi'an Jiaotong University will be enrolled into the study. There will be five groups to be observed. Four groups are taking tenofovir to prevent intrauterine infection during pregnancy. One group is not taking any anti-HBV virus treatments.The clinical value and effectiveness of tenofovir on blocking HBV intrauterine infection will be evaluated; The HBV-DNA infection status of placenta tissue will be checked by quantitative Polymerase Chain Reaction (PCR) to assess the changes of HBV-DNA of placenta after treating with tenofovir and explore the mechanism of tenofovir blocking HBV intrauterine infection. The safety of Tenofovir will be assessed as well.

ELIGIBILITY:
Inclusion Criteria:

* pregnancy patients with HBeAg-positive and HBV-DNA≥ 106copies /ml

Exclusion Criteria:

* pregnancy patients with HBeAg-negative or HBV-DNA<106copies /ml

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: pregnant women with HBeAg-positive and HBV-DNA>106copies/ml from the out-patient department of First Affiliated Hospital of Xi'an Jiaotong University
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-03; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
deoxyribonucleic acid of Hepatitis B Virus (HBV-DNA) in serum | up to 1 year
  Check HBV-DNA in serum by ELISA in pregnant women. The measure unit is copies/mL
deoxyribonucleic acid of Hepatitis B Virus (HBV-DNA) in serum | up to 1 year
  Check HBV-DNA in serum by quantitative PCR in pregnant women. The measure unit is copies/mL

SECONDARY OUTCOMES:
the concentration of Interleukin 2 (IL-2) | up to 1 year
  the concentration of Interleukin 2 (IL-2)in serum of pregnant women, U/mL
interferon-γ (IFN-γ) | up to 1 year
  the concentration of interferon-γ (IFN-γ) in serum of pregnant women,U/mL
Interleukin 4 (IL-4) | up to 1 year
  the concentration of Interleukin 4 (IL-4)in serum of pregnant women, U/mL
Interleukin 6 (IL-6) | up to 1 year
  the concentration of Interleukin 6 (IL-6)in serum of pregnant women,U/mL
T cell ratio | up to 1 year
  T cell ratio in serum is measured by follow cytometry in pregnant women
HBV-DNA of babies | when the baby is 7-month-old
  Check HBV-DNA by ELISA and quantitative PCR. The measure unit is copies/mL. All babies who used tenofovir will be tested when he is 7-month-old, in order to make sure whether they have infection during pregnant period.
hepatitis B e-antigen (HBeAg) | up to 1 year
  check HBeAg in serum of pregnant women.the measure unit is PEIU/mL
HBV-DNA in placenta tissue | the date of delivery
  Check HBV-DNA of placenta tissue by quantitative PCR. The measure unit is copies/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Guiqin Bai, M.D.;Ph.D., Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao F, Zhang WT, Lin YY, Wang WM, Xu N, Bai GQ. Early Start Of Tenofovir Treatment Achieves Better Viral Suppression In Pregnant Women With A High HBV Viral Load: A Real-World Prospective Study. Infect Drug Resist. 2019 Nov 7;12:3475-3484. doi: 10.2147/IDR.S228982. eCollection 2019. PMID 31807036